CLINICAL TRIAL: NCT00089661
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Evaluate AMG 162 in the Treatment of Bone Loss in Subjects Undergoing Aromatase Inhibitor Therapy for Non-metastatic Breast Cancer
Brief Title: AMG 162 in the Treatment of Bone Loss in Subjects Undergoing Aromatase Inhibitor Therapy for Non-metastatic Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20040135
Record Dates: First submitted 2004-08-09; First posted 2004-08-11 (Estimated); Results first posted 2010-01-26 (Estimated); Last update posted 2018-10-17 (Actual); Status verified 2018-09

CONDITIONS: Breast Cancer; Low Bone Mineral Density; Osteopenia
Keywords: Breast Cancer; Bone loss associated with Aromatase Inhibitor therapy (AIT) for non-metastatic BC; osteopenia; Low bone density
MeSH Terms: conditions — Breast Neoplasms; Bone Diseases, Metabolic | interventions — Denosumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- AMG 162 / Denosumab (Experimental)
  Interventions: Drug: AMG 162 / Denosumab
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — 60 mg (1.0 mL) administered subcutaneously every six months, beginning on Study Day 1, for a total treatment period of 24 months
  Arms: Placebo
Drug: AMG 162 / Denosumab — 60 mg (1.0 mL) administered subcutaneously every six months, beginning on Study Day 1, for a total treatment period of 24 months
  Arms: AMG 162 / Denosumab

SUMMARY:
The purpose of this trial is to evaluate AMG 162 in the treatment of bone loss in subjects undergoing Aromatase Inhibitor Therapy for Non-metastatic Breast Cancer.

ELIGIBILITY:
* Histologically or cytologically confirmed adenocarcinoma of the breast
* Subjects with early stage disease who are estrogen receptor positive and who have completed their treatment pathway (surgery, chemo-therapy, radiation, and/or hormone therapy) and are currently on or will initiate aromatase inhibitor therapy, and are expected to stay on aromatase inhibitor therapy for the duration of the 24-month study
* All treatment pathway must be completed ≥ 4 weeks prior to study entry, and all acute toxic effect of any above therapy must be resolved to ≤ Grade 1 by National Cancer Institution (NCI) Common Terminology Criteria for Adverse Events (CTCAE)
* Female > 18 years of age
* ECOG Performance status 0 and 1
* Lumbar spine, total hip or femoral neck BMD equivalent to a t-score classification of -1.0 to -2.5
* Subject is willing and able to provide signed consent before any study-specific procedure

Other criteria also apply.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Actual)
Dates: Start 2004-10-01 (Actual); Primary Completion 2007-05-11 (Actual); Study Completion 2009-05-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Background] Ellis GK, Bone HG, Chlebowski R, Paul D, Spadafora S, Fan M, Kim D. Effect of denosumab on bone mineral density in women receiving adjuvant aromatase inhibitors for non-metastatic breast cancer: subgroup analyses of a phase 3 study. Breast Cancer Res Treat. 2009 Nov;118(1):81-7. doi: 10.1007/s10549-009-0352-y. Epub 2009 Mar 24. PMID 19308727
- [Background] Ellis GK, Bone HG, Chlebowski R, Paul D, Spadafora S, Smith J, Fan M, Jun S. Randomized trial of denosumab in patients receiving adjuvant aromatase inhibitors for nonmetastatic breast cancer. J Clin Oncol. 2008 Oct 20;26(30):4875-82. doi: 10.1200/JCO.2008.16.3832. Epub 2008 Aug 25. PMID 18725648
- [Derived] Adams A, Jakob T, Huth A, Monsef I, Ernst M, Kopp M, Caro-Valenzuela J, Wockel A, Skoetz N. Bone-modifying agents for reducing bone loss in women with early and locally advanced breast cancer: a network meta-analysis. Cochrane Database Syst Rev. 2024 Jul 9;7(7):CD013451. doi: 10.1002/14651858.CD013451.pub2. PMID 38979716
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com
- See also: Notice regarding posted summaries of trial results — http://download.veritasmedicine.com/REGFILES/amgen/Amgen_results_disclaimer.pdf

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Denosumab 60 mg Q6M | Placebo
Started | 127 | 125
Completed | 106 | 99
Not Completed | 21 | 26
Not completed — Adverse Event | 0 | 2
Not completed — Death | 1 | 0
Not completed — Lost to Follow-up | 0 | 3
Not completed — Withdrawal by Subject | 11 | 9
Not completed — Disease progression | 1 | 3
Not completed — Ineligibility determined | 4 | 4
Not completed — Noncompliance | 2 | 4
Not completed — Other | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Denosumab 60 mg Q6M | Placebo | Total
Number analyzed (Participants) | 127 | 125 | 252
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.2 (8.9) | 59.7 (9.7) | 59.5 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 127 | 125 | 252
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Lumbar Spine Bone Mineral Density Percent Change From Baseline at Month 12
Description: Bone Mineral Density Assessed by Dual Energy X-Ray Absorptiometry.
Time Frame: 12 months
Population: Subjects with non-missing baseline and >= 1 non-missing post-baseline evaluation. Using Last Observation Carried Forward as imputation.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change from Baseline
Arm/Group | Denosumab 60 mg Q6M | Placebo
Number analyzed (Participants) | 123 | 122
Percent Change from Baseline | 4.8 [4.3 to 5.4] | -.7 [-1.3 to -.1]
Statistical Analysis 1: Comparison: Denosumab 60 mg Q6M vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = 5.5, 95% CI [4.8 to 6.3]

2. Secondary Outcome: Lumbar Spine Bone Mineral Density Percent Change From Baseline at Month 6
Description: Bone Mineral Density Assessed by Dual Energy X-Ray Absorptiometry.
Time Frame: 6 months
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change from Baseline
Arm/Group | Denosumab 60 mg Q6M | Placebo
Number analyzed (Participants) | 123 | 122
Percent Change from Baseline | 3.7 [3.2 to 4.2] | -.6 [-1.1 to -.1]

3. Secondary Outcome: Total Hip Bone Mineral Density Percent Change From Baseline at Month 12
Description: Bone Mineral Density Assessed by Dual Energy X-Ray Absorptiometry.
Time Frame: 12 months
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change from Baseline
Arm/Group | Denosumab 60 mg Q6M | Placebo
Number analyzed (Participants) | 123 | 122
Percent Change from Baseline | 3.1 [2.6 to 3.5] | -.7 [-1.1 to -.2]

4. Secondary Outcome: Total Hip Bone Mineral Density Percent Change From Baseline at Month 6
Description: Bone Mineral Density Assessed by Dual Energy X-Ray Absorptiometry.
Time Frame: 6 months
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change from Baseline
Arm/Group | Denosumab 60 mg Q6M | Placebo
Number analyzed (Participants) | 123 | 122
Percent Change from Baseline | 2.3 [1.9 to 2.8] | -.4 [-.8 to .1]

5. Secondary Outcome: Femoral Neck Bone Mineral Density Percent Change From Baseline at Month 12
Description: Bone Mineral Density Assessed by Dual Energy X-Ray Absorptiometry.
Time Frame: 12 months
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change from Baseline
Arm/Group | Denosumab 60 mg Q6M | Placebo
Number analyzed (Participants) | 123 | 122
Percent Change from Baseline | 1.9 [1.1 to 2.6] | -.6 [-1.4 to .2]

6. Secondary Outcome: Femoral Neck Bone Mineral Density Percent Change From Baseline at Month 6
Description: Bone Mineral Density Assessed by Dual Energy X-Ray Absorptiometry.
Time Frame: 6 months
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change from Baseline
Arm/Group | Denosumab 60 mg Q6M | Placebo
Number analyzed (Participants) | 123 | 122
Percent Change from Baseline | 1.2 [.5 to 1.9] | -.9 [-1.6 to -.2]

ADVERSE EVENTS:
Arm/Group | Placebo | Denosumab 60 mg Q6M
Serious Adverse Events (participants affected / at risk) | 11/120 | 19/129
Other Adverse Events (participants affected / at risk) | 108/120 | 117/129
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=120) | Denosumab 60 mg Q6M (N=129)
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0
Atrioventricular block second degree (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 1 | 0
Goitre (Endocrine disorders) | 1 | 0
Colitis ischaemic (Gastrointestinal disorders) | 0 | 1
Diverticulum (Gastrointestinal disorders) | 0 | 1
Faecaloma (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Large intestine perforation (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Pelvic mass (General disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 1
Cholelithiasis (Hepatobiliary disorders) | 2 | 0
Cellulitis (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 1
Labyrinthitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 1
Incisional hernia (Injury, poisoning and procedural complications) | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 2
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Benign ovarian tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 1
Rectocele (Reproductive system and breast disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=120) | Denosumab 60 mg Q6M (N=129)
Constipation (Gastrointestinal disorders) | 11 | 15
Diarrhoea (Gastrointestinal disorders) | 9 | 5
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 8 | 2
Nausea (Gastrointestinal disorders) | 11 | 10
Vomiting (Gastrointestinal disorders) | 6 | 8
Fatigue (General disorders) | 17 | 17
Oedema peripheral (General disorders) | 5 | 8
Bronchitis (Infections and infestations) | 7 | 5
Sinusitis (Infections and infestations) | 4 | 9
Upper respiratory tract infection (Infections and infestations) | 6 | 10
Urinary tract infection (Infections and infestations) | 5 | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 30 | 31
Arthritis (Musculoskeletal and connective tissue disorders) | 6 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 15 | 18
Bone pain (Musculoskeletal and connective tissue disorders) | 8 | 5
Muscle spasms (Musculoskeletal and connective tissue disorders) | 6 | 7
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 6 | 7
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 11
Pain in extremity (Musculoskeletal and connective tissue disorders) | 14 | 19
Shoulder pain (Musculoskeletal and connective tissue disorders) | 4 | 11
Headache (Nervous system disorders) | 9 | 11
Hypoaesthesia (Nervous system disorders) | 4 | 7
Anxiety (Psychiatric disorders) | 6 | 8
Depression (Psychiatric disorders) | 11 | 7
Insomnia (Psychiatric disorders) | 14 | 12
Breast pain (Reproductive system and breast disorders) | 6 | 3
Vulvovaginal dryness (Reproductive system and breast disorders) | 3 | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 13
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 7
Rash (Skin and subcutaneous tissue disorders) | 6 | 10
Hot flush (Vascular disorders) | 8 | 7
Hypertension (Vascular disorders) | 7 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multi-center studies, the investigator agrees not to publish any results before the first multi-center publication.